CLINICAL TRIAL: NCT00391118
Title: A Randomized, Phase 2, Placebo-Controlled, Double-Blinded Study With and Without Enzastaurin in Combination With Paclitaxel and Carboplatin as First-Line Treatment, Followed by Maintenance Treatment in Advanced Ovarian Cancer
Brief Title: Comparing Two Treatments for Ovarian Cancer: Standard Chemotherapy Plus Enzastaurin, or Placebo ("Sugar Pill")
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10708; H6Q-MC-S019 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Cancer; Fallopian Tube Neoplasms; Peritoneal Neoplasm
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — enzastaurin; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Part A) (Experimental): Enzastaurin: 1125 milligram (mg) loading dose then 500 mg oral tablet, daily for six 21-day cycles or up to 3 years
  Carboplatin: Area under the concentration time curve (AUC) 5 intravenous (IV), every (q) 21 days for six 21-day cycles
  Paclitaxel:175 milligrams/square meter (mg/m²) IV, q21 days for six 21-day cycles
  Interventions: Drug: enzastaurin; Drug: carboplatin; Drug: paclitaxel
- B (Part B) (Placebo Comparator): Carboplatin: AUC5 IV, q21 days for six 21-day cycles
  Paclitaxel: 175 mg/m², IV, q21 days for six 21-day cycles
  Placebo: oral tablet
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: placebo

INTERVENTIONS:
Drug: enzastaurin
  Other Names: LY317615
  Arms: A (Part A)
Drug: carboplatin
Drug: paclitaxel
Drug: placebo
  Arms: B (Part B)

SUMMARY:
Participants with ovarian cancer usually get the drugs carboplatin and paclitaxel as initial treatment. In many participants the tumor will shrink, or even disappear, after treatment with these drugs. But, unfortunately, the tumor will grow again in many participants. This trial will try to address the question: Can we delay the time till the tumor grows again by adding a 3rd drug to the standard therapy? To answer this question, participants will, by chance, either get the experimental drug enzastaurin or a "dummy pill" (placebo) during the chemotherapy and for up to 3 years after chemotherapy. Participants and physicians will not know if a participant gets enzastaurin or placebo (double-blinded trial). After a predefined time, the treatment will be uncovered, and the number of participants with tumor growth at a specific time point will be compared between the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have specific stages of disease, known as Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) stages IIB, IIC, III or IV
* Organ functions (blood, renal, liver, cardiac) must meet specific requirements.
* Participants who could become pregnant must take care not to become pregnant during the study participation and for 6 months after study discontinuation
* Participants must give written consent for study participation.

Exclusion Criteria:

* Participants received any experimental drug within the last 30 days.
* Participants received any prior chemotherapy or other drug therapy for the current disease.
* Participants receive any other treatment for the cancer during study participation.
* Participants are unable to discontinue concurrent administration of carbamazepine, phenobarbital, or phenytoin.
* Participants are pregnant, breast feeding, or not using adequate contraceptive methods to prevent pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wiesbaden
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivanovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1: Unblinded, single cohort safety lead-in of enzastaurin (enz) with paclitaxel (pac)/carboplatin (carb). Part 2: Randomized, double-blind, placebo-controlled trial consisting of: Baseline, Chemotherapy (start of study drug to discontinuation of pac and carb), Maintenance (day chemotherapy ends to study completion), Follow-up (up to 3 years).
Groups:
- Part 1 - Modified Regimen A: Enzastaurin: 1125 milligrams (mg) loading dose on Cycle 1 Day 4 then 500 mg oral tablet, daily (QD), for six 21-day cycles on subsequent days of chemotherapy
  Carboplatin: Area under the concentration time curve (AUC)5 intravenous (IV), every (q) 21 days, for six 21-day cycles of chemotherapy
  Paclitaxel: 175 milligrams/square meter (mg/m²), IV, q21 days, for six 21-day cycles of chemotherapy
- Part 2 - Regimen A: Enzastaurin: 1125 mg loading dose then 500 mg oral tablet on subsequent days, QD, for six 21-day cycles of chemotherapy and maintenance therapy up to 2 years
  Carboplatin: AUC5, IV, q21 days, for six 21-day cycles of chemotherapy
  Paclitaxel: 175 mg/m², IV, q21 days, for six 21-day cycles of chemotherapy
- Part 2 - Regimen B: Carboplatin: AUC5, IV, q21 days for six 21-day cycles of chemotherapy
  Paclitaxel: 175 mg/m², IV, q21 days for six 21-day cycles of chemotherapy
  Placebo: oral tablet, QD of chemotherapy and maintenance therapy up to 2 years
Period: Overall Study
Arm/Group | Part 1 - Modified Regimen A | Part 2 - Regimen A | Part 2 - Regimen B
Started | 11 | 69 | 73
Received ≥1 Dose of Assigned Study Drug | 11 | 67 | 72
Completed | 0 | 14 | 15
Not Completed | 11 | 55 | 58
Not completed — Adverse Event | 3 | 10 | 7
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 9 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Physician Decision | 0 | 3 | 0
Not completed — Protocol Entry Criteria Not Met | 0 | 3 | 1
Not completed — Progressive Disease | 7 | 26 | 43
Not completed — Sponsor Decision | 0 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1: All enrolled participants Part 2: All randomized participants
Groups:
- Part 1 - Modified Regimen A: Enzastaurin: 1125 mg loading dose on Cycle 1 Day 4 then 500 mg oral tablet, QD, for six 21-day cycles on subsequent days of chemotherapy
  Carboplatin: AUC5, IV, q21 days, for six 21-day cycles of chemotherapy
  Paclitaxel: 175 mg/m², IV, q21 days, for six 21-day cycles of chemotherapy
- Part 2 - Regimen A: Enzastaurin: 1125 mg loading dose then 500 mg oral tablet, QD, for up to six 21-day cycles on subsequent days of chemotherapy and maintenance therapy up to 2 years
  Carboplatin: AUC5, IV, q21 days, for up to six 21-day cycles of chemotherapy
  Paclitaxel: 175 mg/m², IV, q21 days, for up to six 21-day cycles of chemotherapy
- Part 2 - Regimen B: Carboplatin: AUC5 IV, q21 days, for up to six 21-day cycles of chemotherapy
  Paclitaxel: 175 mg/m², IV, q21 days, for up to six 21-day cycles of chemotherapy
  Placebo: oral tablet, QD, of chemotherapy and maintenance therapy up to 2 years
- Total: Total of all reporting groups
Arm/Group | Part 1 - Modified Regimen A | Part 2 - Regimen A | Part 2 - Regimen B | Total
Number analyzed (Participants) | 11 | 69 | 73 | 153
Age, Continuous [Median (Full Range); unit: years] | 52.4 [41.4 to 74.4] | 55.3 [27.6 to 73.9] | 53.4 [19.6 to 78.8] | 54.90 [19.6 to 78.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 69 | 73 | 153
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 68 | 72 | 151
  East Asian | 0 | 1 | 0 | 1
  West Asian (Indian sub-continent) | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 5 | 14 | 13 | 32
  Poland | 0 | 7 | 7 | 14
  Spain | 0 | 3 | 8 | 11
  Russia | 0 | 17 | 20 | 37
  Germany | 6 | 28 | 25 | 59

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Progression-Free Survival (PFS)
Description: PFS was defined as time from date of randomization to first date of determined progressive disease (PD) or death from any cause. PD defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) and Gynecological Cancer Intergroup (GCIG) criteria. RECIST: ≥20% increase in sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since treatment started or appearance of ≥ 1new lesions and/or unequivocal progression of existing non-target lesions. GCIG: Cancer Antigen-125 (CA-125) serum ≥2 times upper limit of normal (ULN) for those in normal range or nadir for participants who never achieved normal range. Participants not known to have died and did not have PD were censored at last progression-free assessment. Those who received subsequent systemic anticancer therapy (after study drug discontinued) prior to determined PD or death, were censored at date of last progression-free disease assessment prior to post-discontinuation chemotherapy.
Time Frame: Randomization up to date of PD or death (up to 28.6 months)
Population: All randomized participants from Part 2 group. Participants censored for Part 2: Regimen A=38, Regimen B=35. Per protocol, Part 1 was not included as it is an open-label safety lead-in portion with PK characterization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2 - Regimen A | Part 2 - Regimen B
Number analyzed (Participants) | 69 | 73
months | 18.9 [13.8 to NA] — Upper level of confidence interval not calculated due to high censoring. | 15.2 [11.0 to 18.9]

2. Secondary Outcome: Part 2: Percentage of Participants With PFS at 2 Years
Description: PFS was defined as time from date of randomization to first date of determined PD or death from any cause. PD defined using RECIST v1.0 and GCIG criteria. RECIST v1.0: as ≥20% increase in sum of LD of target lesions taking as reference the smallest sum LD recorded since treatment started or appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. GCIG: CA-125 serum ≥2 times ULN for those in normal range or nadir (the lowest value of blood counts after chemotherapy) for participants who never achieved normal range. Participants not known to have died and did not have PD were censored at last progression-free assessment. Those who received subsequent systemic anticancer therapy (after study drug discontinued) prior to determined PD or death, were censored at date of last progression-free disease assessment prior to post-discontinuation chemotherapy.
Time Frame: Randomization to measured PD evaluated at 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2 - Regimen B: Carboplatin: AUC5, IV, q21 days, for up to six 21-day cycles of chemotherapy
  Paclitaxel: 175 mg/m², IV, q21 days, for up to six 21-day cycles of chemotherapy
  Placebo: oral tablet, QD, of chemotherapy and maintenance therapy up to 2 years
Arm/Group | Part 2 - Regimen A | Part 2 - Regimen B
Number analyzed (Participants) | 69 | 73
percentage of participants | 35.2 [20.4 to 50.4] | 28.2 [15.7 to 42.2]

3. Secondary Outcome: Part 2: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: ORR was the percentage of participants with a CR or PR using RECIST v1.0 and CA-125 GCIG criteria. RECIST v1.0: CR was defined as the disappearance of all tumors. PR was defined ≥30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD or complete disappearance of target lesions, with persistence (but not worsening) of ≥1 nontarget lesions and appearance of no new lesions. GCIG: CA-125 serum ≥2 times above ULN for those in normal range or nadir for participants who never achieved normal range. ORR calculated as: (CR + PR) / (total number of participants qualified for tumor response analysis per arm) * 100.
Time Frame: Randomization to PD or death from any cause (up to 28.6 months)
Population: All randomized participants from Part 2 group, who were evaluated for tumor response. Per protocol, Part 1 was not included as it is an open-label safety lead-in portion with PK characterization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 - Regimen A | Part 2 - Regimen B
Number analyzed (Participants) | 14 | 18
percentage of participants | 42.9 [17.7 to 71.1] | 38.9 [17.3 to 64.3]

4. Secondary Outcome: Part 2: Percentage of Participants With CR or PR or Stable Disease (SD) (Rate of Response)
Description: Rate of response was defined using RECIST v1.0 and CA-125 GCIG criteria. RECIST v1.0: CR was defined as the disappearance of all target lesions. PR was defined ≥30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD or complete disappearance of target lesions, with persistence (but not worsening) of ≥1 nontarget lesions and appearance of no new lesions. SD was defined as small changes that did not meet the above criteria. PD was defined as having a ≥20% increase in the sum of the LD of target lesions. GCIG: CA-125 serum ≥2 times above ULN for those in normal range or nadir for participants who never achieved normal range. Rate of response calculated as: (CR + PR + SD)/(total number of participants qualified for tumor response analysis per arm) *100.
Time Frame: Randomization to PD or death from any cause (up to 28.6 months)
Population: All randomized participants from Part 2 group, who qualified for tumor response analysis. Per protocol, Part 1 was not included as it is an open-label safety lead-in portion with PK characterization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 - Regimen A | Part 2 - Regimen B
Number analyzed (Participants) | 14 | 18
percentage of participants
  CR | 7.1 [0.2 to 33.9] | 22.2 [6.4 to 47.6]
  PR | 35.7 [12.8 to 64.9] | 16.7 [3.6 to 41.4]
  SD | 42.9 [17.7 to 71.1] | 50.0 [26.0 to 74.0]

5. Secondary Outcome: Part 2: Translational Research: PFS Based on Protein Expression (PE) (To Assess Biological Markers in Tumors That Could Indicate Who Could Benefit From Enzastaurin Treatment)
Description: PE measured using Immunohistochemistry (IHC) assay, scored 0 (negative, no staining) to 3+ (brightest staining). IHC H-scores for protein biomarkers (PKCβ2, PTEN, pCREB, pGSK3b, pS6) calculated as: [1*(percentage of cells stained [PCS] as 1+)]+[2*(PCS as 2+)]+[3*(PCS as 3+)]. High PE: ≥marker threshold value and Low PE: <marker threshold value. PFS: date of randomization to PD or death. PD defined using RECIST v1.0 and GCIG criteria. RECIST: ≥20% increase in sum of LD of target lesions taking as references smallest sum LD recorded since treatment started or appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. GCIG: CA-125 serum ≥2 times ULN for those in normal range or nadir for those who never achieved normal range. Per protocol, Part 1 was not included as it is an open-label safety lead-in portion with PK characterization.
Time Frame: Randomization up to date of PD or death (up to 28.6 months)
Population: All randomized participants (Pts) from Part 2 group. Pts censored: Regimens A/B (A/B)-High (H), Low (L) Expression: PKCβ2 Cytoplasm (Cyto) (H4/5,L26/22), PTEN Cyto (H24/24, L6/3), PTEN Membrane (H9/8, L21/19), PTEN Nucleus (H13/6, L17/21), pCREB Nucleus (H14/10, L16/17), pGSK3b Cyto (H7/3, L22/23), pS6 Cyto (H21/18, L9/9).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2 - Regimen A | Part 2 - Regimen B
Number analyzed (Participants) | 56 | 55
months
  PKCβ2 Cytoplasm High Expression (H≥115): number analyzed (Participants) | 7 | 14
  PKCβ2 Cytoplasm High Expression (H≥115) | 18.9 [12.8 to NA] — Upper limit of Confidence Interval was not reached. | 10.4 [8.0 to 18.0]
  PKCβ2 Cytoplasm Low Expression (H<115): number analyzed (Participants) | 49 | 41
  PKCβ2 Cytoplasm Low Expression (H<115) | 19.1 [12.1 to NA] — Upper limit of Confidence Interval was not reached. | 18.2 [13.3 to NA] — Upper limit of Confidence Interval was not reached.
  PTEN Cytoplasm High Expression (H≥50): number analyzed (Participants) | 46 | 41
  PTEN Cytoplasm High Expression (H≥50) | 18.9 [12.1 to 19.6] | 18.2 [16.8 to NA] — Upper limit of Confidence Interval was not reached.
  PTEN Cytoplasm Low Expression (H<50): number analyzed (Participants) | 10 | 14
  PTEN Cytoplasm Low Expression (H<50) | NA [14.0 to NA] — Median not calculated due to high rate of censoring and Upper limit of Confidence Interval was not reached. | 10.4 [8.2 to 13.3]
  PTEN Membrane High Expression (H≥15): number analyzed (Participants) | 20 | 11
  PTEN Membrane High Expression (H≥15) | 18.4 [10.3 to 19.6] | NA [11.7 to NA] — Median not calculated due to high rate of censoring and Upper limit of Confidence Interval was not reached.
  PTEN Membrane Low Expression (H<15): number analyzed (Participants) | 36 | 44
  PTEN Membrane Low Expression (H<15) | 19.1 [10.9 to NA] — Upper limit of Confidence Interval was not reached. | 14.7 [11.0 to 18.0]
  PTEN Nucleus High Expression (H≥12): number analyzed (Participants) | 19 | 14
  PTEN Nucleus High Expression (H≥12) | NA [13.9 to NA] — Median not calculated due to high rate of censoring and Upper limit of Confidence Interval was not reached. | 16.8 [8.7 to NA] — Upper limit of Confidence Interval was not reached.
  PTEN Nucleus Low Expression (H<12): number analyzed (Participants) | 37 | 41
  PTEN Nucleus Low Expression (H<12) | 18.4 [10.3 to 19.6] | 16.9 [11.7 to NA] — Upper limit of Confidence Interval was not reached.
  pCREB Nucleus High Expression (H≥217): number analyzed (Participants) | 21 | 20
  pCREB Nucleus High Expression (H≥217) | 19.6 [18.4 to NA] — Upper limit of Confidence Interval was not reached. | 13.2 [9.2 to NA] — Upper limit of Confidence Interval was not reached.
  pCREB Nucleus Low Expression (H<217): number analyzed (Participants) | 34 | 33
  pCREB Nucleus Low Expression (H<217) | 14.0 [10.5 to NA] — Upper limit of Confidence Interval was not reached. | 18.2 [12.1 to NA] — Upper limit of Confidence Interval was not reached.
  pGSK3b Cytoplasm High Expression (H≥160): number analyzed (Participants) | 10 | 7
  pGSK3b Cytoplasm High Expression (H≥160) | NA [18.9 to NA] — Median not calculated due to high rate of censoring and Upper limit of Confidence Interval was not reached. | 14.5 [11.7 to NA] — Upper limit of Confidence Interval was not reached.
  pGSK3b Cytoplasm Low Expression (H<160): number analyzed (Participants) | 45 | 46
  pGSK3b Cytoplasm Low Expression (H<160) | 14.0 [10.3 to 19.6] | 17.4 [11.0 to NA] — Upper limit of Confidence Interval was not reached.
  pS6 Cytoplasm High Expression (H≥105): number analyzed (Participants) | 35 | 35
  pS6 Cytoplasm High Expression (H≥105) | 19.6 [18.4 to NA] — Upper limit of Confidence Interval was not reached. | 18.0 [11.7 to NA] — Upper limit of Confidence Interval was not reached.
  pS6 Cytoplasm Low Expression (H<105): number analyzed (Participants) | 21 | 19
  pS6 Cytoplasm Low Expression (H<105) | 11.5 [9.9 to 19.6] | 17.4 [11.0 to NA] — Upper limit of Confidence Interval was not reached.

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Other Non-Serious Adverse Events (AEs) and the Number of Participants Who Died (To Compare the Safety of the 2 Treatments)
Description: Clinically significant events were defined as SAEs and other non-serious AEs regardless of causality. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module. The number of participants SAEs, other non-serious AEs, and those who died due to PD are included.
Time Frame: Randomization up to 28.6 months
Population: All enrolled (Part 1) and all randomized (Part 2) participants who received at least 1 dose of study drug according to the treatment to which the participants were assigned.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 - Modified Regimen A: Enzastaurin: 1125 mg loading dose on Cycle 1 Day 4 then 500 mg oral tablet, QD, for six 21-day cycles on subsequent days of chemotherapy
  Carboplatin: AUC5, IV, q 21 days, for six 21-day cycles of chemotherapy
  Paclitaxel: 175 mg/m², IV, q21 days, for six 21-day cycles of chemotherapy
Arm/Group | Part 1 - Modified Regimen A | Part 2 - Regimen A | Part 2 - Regimen B
Number analyzed (Participants) | 11 | 67 | 72
Participants
  SAEs | 7 | 26 | 20
  Non-Serious AEs | 11 | 60 | 56
  Died | 0 | 3 | 0

7. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) for Carboplatin With and Without Enzastaurin for Part 1 of Study
Time Frame: Cycle 1 Day 1 (carb) and Cycle 2 Day 1 (carb + enz); carb 0.25 hours (h) (prior to infusion), 0.5, 1, 2, 3, 5, and 21h after start of infusion
Population: All enrolled participants with measurable Cmax in Part 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Part 1 - Modified Regimen A
Number analyzed (Participants) | 10
micrograms/milliliter (µg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 9
  Cycle 1 Day 1 | 11.1 (21)
  Cycle 2 Day 1 | 10.8 (13)

8. Secondary Outcome: PK: Cmax for Paclitaxel With and Without Enzastaurin for Part 1 of Study
Time Frame: Cycle 1 Day 1 (pac) and Cycle 2 Day 1 (pac + enz); pac 1, 2, 3h (immediately after stopping infusion), 3.25, 3.5, 4, 5, 6, 8, 24, and 30h after start of infusion
Population: All enrolled participants with measurable Cmax for pac in Part 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Part 1 - Modified Regimen A
Number analyzed (Participants) | 8
nanograms/milliliter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 7
  Cycle 1 Day 1 | 3580 (43)
  Cycle 2 Day 1 | 3670 (33)

9. Secondary Outcome: PK: AUC From Time 0 to Infinity (AUC0-∞) for Carboplatin With and Without Enzastaurin for Part 1 of Study
Time Frame: Cycle 1 Day 1 (carb) and Cycle 2 Day 1 (carb + enz); carb at 0.25h (prior to infusion), 0.5, 1, 2, 3, 5, and 21h after start of infusion
Population: All enrolled participants with measurable AUC0-∞ in Part 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams*minute/milliliter (mg*min/mL
Arm/Group | Part 1 - Modified Regimen A
Number analyzed (Participants) | 10
milligrams*minute/milliliter (mg*min/mL
  Cycle 1 Day 1: number analyzed (Participants) | 9
  Cycle 1 Day 1 | 3.32 (10)
  Cycle 2 Day 1 | 3.80 (16)

10. Secondary Outcome: PK: AUC0-∞ for Paclitaxel With and Without Enzastaurin for Part 1 of Study
Time Frame: Cycle 1 Day 1 (pac) and Cycle 2 Day 1 (pac + enz); pac at 1, 2, 3h (immediately after stopping infusion), 3.25, 3.5, 4, 5, 6, 8, 24, and 30h after start of infusion
Population: All enrolled participants with measurable AUC0-∞ in Part 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 1 - Modified Regimen A
Number analyzed (Participants) | 8
ng*h/mL
  Cycle 1 Day 1: number analyzed (Participants) | 7
  Cycle 1 Day 1 | 12000 (24)
  Cycle 2 Day 1 | 14400 (23)

11. Secondary Outcome: PK: Cmax at Steady State (Cmax,ss) for Part 1 of Study
Description: Cmax,ss for enzastaurin, its metabolite LSN326020 (LY326020) and total analytes are reported.
Time Frame: Cycle 1 Day 21 (enz) and Cycle 2 Day 1 (carb + pac + enz) at pre-dose, 2, 4, 6, 8 and 24h after the enz dose
Population: All enrolled participants with measurable Cmax,ss in Part 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Part 1 - Modified Regimen A
Number analyzed (Participants) | 9
nmol/L
  Enzastaurin Cycle 1 Day 21 | 1230 (110)
  Enzastaurin Cycle 2 Day 1 | 935 (80)
  LSN326020 Cycle 1 Day 21 | 890 (58)
  LSN326020 Cycle 2 Day1 | 814 (30)
  Total Analyte Cycle 1 Day 21 | 2190 (81)
  Total Analyte Cycle 2 Day 1 | 1640 (57)

12. Secondary Outcome: PK: AUC During the Dosing Interval at Steady State (AUCτ,ss) for Part 2 of Study
Description: AUCτ,ss for enzastaurin, its metabolite LSN326020 (LY326020), and total analytes are reported.
Time Frame: Cycle 2 Day 1 (carb + pac + enz) at pre-dose, 2, 4, 6, 8 and 24h after the enz dose
Population: All randomized participants with measurable AUCτ,ss in Part 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Part 2 - Regimen A
Number analyzed (Participants) | 23
nmol*h/L
  Enzastaurin | 47100 (95)
  LSN326020 | 55600 (47)
  Total Analyte | 106000 (63)

ADVERSE EVENTS:
Groups:
- Part 1 - Modified Regimen A: Enzastaurin: 1125 mg loading dose on Cycle 1 Day 4, then 500 mg oral tablet, QD, for six 21-day cycles on subsequent days of chemotherapy
  Carboplatin: AUC5, IV, q21 days, for six 21-day cycles
  Paclitaxel: 175 mg/m² IV, q21 days, for six 21-day cycles
- Part 2 - Regimen A: Enzastaurin: 1125 mg loading dose then 500 mg, oral tablets on subsequent days, QD, for six 21-day cycles or up to 2 years
  Carboplatin: AUC5, IV, q 21 days, for six 21-day cycles
  Paclitaxel: 175 mg/m², IV, q21 days, for six 21-day cycles
- Part 2 - Regimen B: Carboplatin: AUC5, IV, q21 days, for six 21-day cycles
  Paclitaxel: 175 mg/m2² IV, q 21 days, six 21 day cycles
  Placebo: oral tablet, QD
Arm/Group | Part 1 - Modified Regimen A | Part 2 - Regimen A | Part 2 - Regimen B
Serious Adverse Events (participants affected / at risk) | 7/11 | 26/67 | 20/72
Other Adverse Events (participants affected / at risk) | 11/11 | 60/67 | 56/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Modified Regimen A (N=11) | Part 2 - Regimen A (N=67) | Part 2 - Regimen B (N=72)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (7) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Keratosis follicular (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal perforation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 2 (10) | 2 (2)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 - Modified Regimen A (N=11) | Part 2 - Regimen A (N=67) | Part 2 - Regimen B (N=72)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 11 (20) | 12 (13)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 10 (18) | 13 (34)
Neutropenia (Blood and lymphatic system disorders) | 6 (16) | 22 (62) | 27 (78)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 4 (5)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 1 (1) | 2 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 15 (27) | 16 (20)
Abdominal pain upper (Gastrointestinal disorders) | 2 (5) | 10 (12) | 6 (7)
Constipation (Gastrointestinal disorders) | 6 (9) | 15 (24) | 22 (34)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 15 (25) | 8 (21)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (5)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (6) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (21) | 30 (77) | 35 (81)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 5 (5) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (11) | 16 (32) | 16 (24)
Asthenia (General disorders) | 0 (0) | 5 (7) | 9 (11)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 7 (21) | 31 (64) | 25 (66)
Mucosal inflammation (General disorders) | 1 (1) | 3 (7) | 6 (12)
Oedema (General disorders) | 0 (0) | 5 (8) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 8 (8)
Pain (General disorders) | 0 (0) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 6 (6) | 3 (3)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (7) | 8 (10)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (14) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 5 (7)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 5 (7) | 3 (4)
Urine colour abnormal (Investigations) | 0 (0) | 4 (4) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 21 (29) | 21 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3) | 7 (17)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 5 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 16 (31) | 15 (28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (9) | 5 (6) | 14 (17)
Dizziness (Nervous system disorders) | 0 (0) | 5 (7) | 6 (6)
Dysgeusia (Nervous system disorders) | 2 (2) | 6 (11) | 12 (14)
Headache (Nervous system disorders) | 2 (2) | 14 (21) | 10 (20)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 5 (6) | 5 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (9) | 24 (29) | 22 (27)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 6 (6) | 4 (4)
Sleep disorder (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (2)
Renal pain (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 41 (41) | 38 (39)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 7 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (11) | 8 (9)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Enterostomy (Surgical and medical procedures) | 1 (2) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (4) | 3 (3) | 6 (10)
Hot flush (Vascular disorders) | 0 (0) | 3 (3) | 5 (5)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
All of the percentages do not add up to 100% because of rounding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days